CLINICAL TRIAL: NCT03322371
Title: Validation of Frontal Limited Lead Electroencephalography (EEG) to Formal Polysomnography (PSG) in the Intensive Care Unit (ICU)
Brief Title: Validation of Frontal EEG to Formal Polysomnography in the ICU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty analyzing PSG data
Sponsor: University of Utah (Other)
Collaborators: Epitel, Inc. (Industry)
Responsible Party: Principal Investigator, Joseph Tonna, Associate Director, ECMO Services, University of Utah
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 87693
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Sleep Deprivation; Sleep
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Health Subjects in Sleep Lab (Other): Adult patients (> 18yrs old) scheduled for a standard of care PSG (sleep study) lasting at least 8 hours for any condition. Patients will undergo simultaneous 2-lead limited EEG recording with experimental device. 2-lead limited electroencephalography recording
  Interventions: Device: 2-lead limited electroencephalography recording
- ICU patients, not sedated or ventilated (Other): Adult ICU patients (> 18yrs old) anticipated to stay in the ICU overnight (minimum 8 hours) with a Glasgow Coma Scale of 13 or greater, not intubated and not sedated. Patients will undergo simultaneous 2-lead limited electroencephalography recording
  Interventions: Device: 2-lead limited electroencephalography recording
- ICU patients, sedated and ventilated (Other): Adult ICU patients (> 18yrs old) who are intubated, sedated, ventilated, and anticipated to stay in the ICU overnight (minimum 8 hours). Patients will undergo simultaneous 2-lead limited electroencephalography recording
  Interventions: Device: 2-lead limited electroencephalography recording

INTERVENTIONS:
Device: 2-lead limited electroencephalography recording — The EEG recording device will be placed in conjunction with the standard formal polysomnography (PSG). The EEG device will remain in place as long as PSG leads are connected to the subject and PSG machine.
  Other Names: Health Subjects in Sleep Lab; ICU patients, not sedated or ventilated; ICU patient, sedated and ventilated

SUMMARY:
The purpose of this study is to compare a 2-lead frontal electroencephalogram recording to a formal polysomnography (PSG) in detecting sleep vs. wake and depth of sleep in both healthy and ICU patients.

DETAILED DESCRIPTION:
Sleep in the intensive care unit (ICU) is poor and not well understood. Formal polysomnography (PSG) is the gold standard measure, but impractical for critical care. The relative influence of environment, illness and interventions on sleep in critically ill patients is therefore essentially unknown. Interventions to improve sleep have been pragmatic and outcomes subjective or indirect, and uninformed. When it is done, formal PSG in critical illness demonstrates fragmented, shortened, interrupted and non-circadian sleep, with environmental noise, light, and frequent physical stimulation causing arousals.

ELIGIBILITY:
Group 1: Healthy Subjects in Sleep Lab:

Inclusion Criteria

* Age 18 or older
* Scheduled for a standard of care polysomnography lasting at least 8 hours for any condition

Exclusion Criteria

* Patient/Legally Authorized Representative declines consent

Group 2: ICU patient, not sedated, not ventilated

Inclusion Criteria

* Age 18 or older
* Anticipated to stay in intensive care unit overnight (minimum 8 hours)
* Glasgow Coma Scale score of 13 or great

Exclusion Criteria:

* Intubated with endotracheal tube
* Sedated (includes sedative drugs such as propofol, Dexmedetomidine, versed infusion above 2mg/hr, ketamine infusion above 0.2 mg/kg/hr).

Group 3: ICU patient, sedated and ventilated

Inclusion Criteria:

* Age 18 or older
* Anticipated to stay in the intensive care unit overnight (minimum 8 hours)
* Intubated, sedated, and ventilated

Exclusion Criteria:

* Presence of traumatic brain injury
* Planned extubation in next 8 hours
* Scheduled to leave the intensive care unit for any reason in the next 8 hours
* Anticipated life expectancy of less than 24 hours
* Electroencephalogram monitoring (current or scheduled in the next 8 hours)
* Hemodynamic instability (defined as: (i) mean arterial pressure <60mmHg for >20 minutes with efforts to raise it or (ii) >2 liter fluid administered in 2h after operating room and anticipating on-going needs for fluid resuscitation or (iii) ICU MD determination of "atypical and profound hemodynamic instability" or (iv) PI determination after evaluation.
* Refractory hypoxemia - defined as Saturation <88% on Sp02 despite efforts to increase it
* Hemorrhage - defined as >500cc chest tube output in 2h and anticipated need of more than 2 units of packed red blood cells in immediate post op period. This does NOT include cell-saver.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Sleep Stage Correlation | Overnight (with a minimum of 960 epochs)
  The correlation of each sleep stage (Wake, NREM1, NREM2, NREM3, REM) as assessed by polysomnography vs. EEG via analysis of 30-second intervals (epochs)

SECONDARY OUTCOMES:
Sleep vs Wake Correlation | Overnight (with a minimum of 960 epochs)
  The correlation of sleep (NREM1, NREM2, NREM3, REM) vs wake as assessed by polysomnography vs. EEG via analysis of 30-second intervals (epochs)

OTHER OUTCOMES:
Sound and Light during Sleep | Overnight (with a minimum of 960 epochs)
  The correlation of sleep stage (Wake, NREM1, NREM2, NREM3, REM) with sound and light levels within the ICU.
Environmental Conditions during Sleep | Overnight (with a minimum of 960 epochs)
  The correlation of sleep stage (Wake, NREM1, NREM2, NREM3, REM) with environmental conditions within the ICU.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Tonna, MD, FAAEM, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States